CLINICAL TRIAL: NCT01055327
Title: Monitoring of Specific Birth Defects Associated With Exposure to Lamotrigine in Pregnancy Through the EUROCAT Network
Brief Title: Birth Defects Associated With Exposure to Lamotrigine in Pregnancy (EUROCAT)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113038
Record Dates: First submitted 2010-01-21; First posted 2010-01-25 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Epilepsy
Keywords: Isolated oral clefts; lamotrigine; EUROCAT; congenital malformations; anti-epileptic drugs
MeSH Terms: conditions — Epilepsy; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infants/foetuses w/malformations registered in EUROCAT network: Pregnancies resulting in foetus/infant with malformation registered through participating registers within the EUROCAT network
  Interventions: Drug: Lamotrigine monotherapy; Drug: No anti-epileptic drug exposure; Drug: Non lamotrigine anti-epileptic drug monotherapy

INTERVENTIONS:
Drug: Lamotrigine monotherapy — Exposure to lamotrigine monotherapy in the first trimester of pregnancy (time period from first day of menstrual period to 12th week of gestation).
Drug: No anti-epileptic drug exposure — No exposure to anti-epileptic drugs in the first trimester of pregnancy (time period from first day of menstrual period to 12th week of gestation).
Drug: Non lamotrigine anti-epileptic drug monotherapy — Exposure to non lamotrigine monotherapy (with or without valproate) during the first trimester of pregnancy (time period from the first day of the menstrual period to the 12th week of gestation)

SUMMARY:
In 2007 a case control study was completed within the EUROCAT European network of congenital anomaly registers to test the hypothesis that first trimester lamotrigine monotherapy exposure is associated with an increased risk of isolated oral clefts. This study found no statistically significant increased risk of oral clefts compared with other defects following lamotrigine exposure in the uterus. The EUROCAT Antiepileptic Drug (AED) Database, established for the original case control study in 2007, will now be expanded to include an additional five to six years worth of data. These data will provide greater power to investigate the risk of isolated oral clefts, specific cleft types and potential associations with additional specific malformation types (e.g. neural tube defects). Data on cases of isolated oral clefts registered between 1993 and 2012 will be extracted from EUROCAT member registers meeting set inclusion criteria (ensuring completeness of outcome and exposure data). The primary comparison group will include all non oral cleft, non chromosomal malformations as the registers do not collect data on non malformed infants. This study will also be powered to include a second control group of chromosomal malformations, very unlikely to be associated with medication exposure. Data on exposure to anti-epileptic drugs (AEDs) during the first trimester of pregnancy will be extracted along with other key covariates including age of mother, history of epilepsy and gestational age of the infant. Primary analyses, using logistic regression, will compare the lamotrigine monotherapy versus no AED use across case and control groups and a secondary analysis will compare lamotrigine monotherapy versus other AED monotherapy (with and without valproate). Data will also be monitored for patterns of lamotrigine exposure across additional specific malformation groups of interest.

ELIGIBILITY:
Inclusion Criteria:

* Individual population-based registers within EUROCAT are eligible to participate if:
* Anti-epileptic drug exposure is recorded for at least 3 per 1000 malformed infants/fetuses (figures below this threshold indicate potential under reporting of medication exposure).
* Specific drug names or complete 7 digit Anatomical Therapeutic Chemical (ATC) classification codes are available for at least 80% of AED exposed infants/fetuses.

Exclusion Criteria:

* As above

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All infants/fetuses with congenital malformations registered on EUROCAT anti-epileptic drug database between 1995 and 2012 (start date depends on date of lamotrigine registration in country of participating register).
  EUROCAT is a European network of population-based congenital anomaly registers for surveillance. EUROCAT surveys 1.5 million births per year covering 29% of births in EU Member States.
  In 2007, 19 population-based congenital malformation registers within EUROCAT participated in an initial study of the association of lamotrigine exposure in pregnancy and the risk of isolated oral clefts. These registries covered at least part of the population of Austria, Belgium, Croatia, Denmark, Finland, France, Germany, Ireland, Italy, Malta, Norway, Poland, Spain, Switzerland and Wales.
  It is anticipated, that if these registers participate in the current study, the study will cover 8 million births and 200,000 congenital malformation registrations between 1995 and 2012.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2009-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Non chromosomal, non monogenic, isolated oral clefts | Retrospective case control study. All isolated oral cleft malformations registered on congenital malformation registers participating in the EUROCAT anti-epileptic drug database will be extracted irrespective of timing of diagnosis pre- or post natally.

SECONDARY OUTCOMES:
Non oral cleft, non chromosomal malformations | Retrospective case control study. All non oral cleft, non chromsomal malformations recorded on congenital malformation registers participating in EUROCAT anti-epileptic drug database extracted irrespective of diagnosis timing pre or post-natal.
All chromosomal malformations | This is a retrospective case control study. All chromosomal malformations recorded on congenital malformation registers participating in the EUROCAT anti-epileptic drug database will be extracted irrespective of timing of diagnosis pre- or post natally.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline